CLINICAL TRIAL: NCT03157661
Title: A Multicentre Cross-sectional Study of the Prevalence of Hypertensive Disease in Patients Presenting for Elective Surgery in the Western Cape
Brief Title: Prevalence of Hypertensive Disease in Patients Presenting for Elective Surgery in the Western Cape, South Africa
Acronym: HASS
Status: Completed | Type: Observational
Sponsor: University of Cape Town (Other)
Responsible Party: Principal Investigator, Dr Marcin Nejthardt, Dr Marcin Nejhardt, University of Cape Town
Other Study IDs: Hypertension and Surgery Study
Record Dates: First submitted 2017-05-15; First posted 2017-05-17 (Actual); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Hypertensive Episode

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single group study: The study population will involve patients presenting for elective surgery, who fulfil inclusion criteria, in all surgical disciplines with elective surgical slates in the main theatre complex, during the period of the study.
  Inclusion Criteria:
  Patients included in the study will be:
  * > 18 years of age
  * Non-cardiac patients
  * Non-obstetric patients
  * Patients receiving general, neuraxial, regional or local/topical anaesthesia for elective surgical intervention

SUMMARY:
Hypertension is a major medical and public health burden throughout the world. It is estimated that 1 in 3 adult South Africans are diagnosed with hypertension, however detailed statistics reflecting the burden of disease are somewhat lacking. The implications and effects of poorly controlled hypertension and its associated co-morbidities are significant and extensive. In South Africa, hypertension is the single most prevalent cardiovascular risk factor and predominant contributor to cardiovascular disease and mortality.

DETAILED DESCRIPTION:
RESEARCH PROBLEM:

Although the diagnosis of hypertension and initiation of treatment is most frequently made in the primary health care setting, the perioperative period provides clinicians with a unique opportunity to identify patients with hypertensive disease, educate patients about the disease, and, if appropriate, initiate appropriate therapy. Furthermore it provides the opportunity to refer patients for further investigation or follow up at peripheral health care centres for ongoing management. The identification and diagnosis of hypertension as well as the effective management thereof is a primary health care target and serves as an efficient health care strategy in reducing long-term cardiovascular morbidity and mortality, as well as the burden of disease associated complications. There are however, a multitude of reasons to investigate and treat persistent hypertension in the perioperative period. The long-term end organ effects are numerous and add significantly to patient morbidity and mortality. Appropriate blood pressure control has an important long term impact on patient outcome. In the acute peri-operative setting the significance of hypertension is however less clear.

AIMS & OBJECTIVES:

Aim of the Study:

The primary aim of the study is to identify and categorise the prevalence of hypertensive disease in adult patients presenting for non-cardiac, non-obstetric elective surgery in all surgical disciplines at 1 tertiary level institution and 6 secondary hospitals over the determined period of the study.

The secondary aims of the study will include the following 1) categorise the degree of hypertensive disease in the study population 2) identify associated target organ damage and associated risk factors 3) determine patient compliance to treatment.

In a sub-study, the primary objective will be to explore the relationship between pre-operative blood pressure measurement and intra-operative hypotension (mean arterial pressure (MAP) < 55mmHg for > 1minute as defined by Walsh et al.

In order to achieve the aims of the study the following objectives will be sought:

Objectives of the Study related to the prevalence of hypertension:

1. Prevalence and degree of hypertensive disease in adult patients presenting for non-cardiac, non-obstetric, elective surgery in all surgical disciplines with elective theatre lists over the period of the study will be determined by measuring and recording preoperative blood pressure during the pre-assessment anaesthetic consultation and/or immediate preoperative period, using an automated oscillometric blood pressure measurement technique. If the blood pressure is noted to be elevated, two additional readings at least 10 minutes apart will be performed. The lowest recorded blood pressure will be used. The study will identify patients with preoperative in hospital blood pressure measurements as follows:

   * SBP<140 mmHg and DBP <90 mmHg
   * SBP<160 mmHg and DBP<100 mmHg
   * SBP<180 mmHg and DBP<110 mmHg without end organ damage
   * SBP<180 mmHg and DBP<110 mmHg with end organ damage
2. Compliance to anti-hypertensive treatment will be assessed using the Morisky Medication Adherence Questionnaire.

Objectives of the sub-study related to the association of pre-operative blood pressure measurement and intra-operative hypotension:

1. Any episodes of low blood pressure defined as a mean arterial pressure of less than 55mmHg will be recorded as well as the cumulative time spend below this threshold.

METHODOLOGY:

Study Design & Data Collection:

This is a prospective quantitative study at one tertiary and six secondary level institutions involving data collected on adult, non-cardiac, non-obstetric patients presenting for elective surgery for a period of one week (from Monday at 7am to Friday at 7pm).

Data is to be collected by the anaesthesiology registrars and consultants providing anaesthetic services to elective patients, in all surgical disciplines, over the one-week period of the study.

Quantitative data will be recorded on a clinical reporting form (CRF) evaluating:

* General demographic information e.g. age, gender, ethnicity
* General medical information e.g. co-morbid conditions, risk factors for hypertension
* Presence of target organ damage which will be assessed by the presence of appropriate electrocardiographic changes, presence of impaired renal function (elevated creatinine) and/or the presence of retinopathy
* General surgical information e.g. indication for surgery and type of surgery

Study Population & Sample Size:

The study population will involve patients presenting for elective non-cardiac, non-obstetric, surgery who are 18 years of age or older and are able to give consent. For the prevalence of hypertension and compliance to treatment part of the study, all patients regardless of the planned anaesthetic technique will be included. For the sub-study, looking at the pre-operative blood pressure and its association with intraoperative hypotension only patients who receive a general or neuraxial anaesthetic will be included. For the sub-study only, this effectively excludes patients who undergo some form of sedation or local block to facilitate their procedures e.g. cataract extraction.

Measurements:

Blood pressure measurements will be performed with an appropriately sized non-invasive blood pressure cuff, using an automated oscillometric method of blood pressure measurement.

Recruitment & Consent:

Participants will be recruited by convenience sampling. All patients compliant with the inclusion criteria will be included in the study. Data obtained will be collected by various anaesthesiology registrars and consultants, and will not include any specific patient information, thus ensuring patient anonymity. Demographic, medical and surgical information is generally routinely available prior to anaesthetic and surgical intervention. Furthermore, blood pressure measurements are routinely performed and documented. Obtained details will be captured on a clinical reporting form and so patient records will not be altered or removed for study purposes. Finally, no additional measurements, tests or investigations will be performed which might place the patient at risk, or discomfort, or impose any additional cost or burden on patient or institutional resources.

Data Management & Analysis:

Data capture forms will be collected and collated. The information will be captured in Excel for further statistical analysis.

Patients will be risk adjusted for:

* Duration of surgery
* Need for blood transfusion intra-operatively
* Pre-operative anaemia
* ASA status
* Functional status
* Major surgery
* Type of anaesthesia (Dependant on sample size)

ETHICAL & LEGAL CONSIDERATIONS:

To ensure complete anonymity, no personal patient information or details will be recorded on the data collection form. As this is an audit, and the researcher will not be involved in delivery of anaesthetic care to the patients in the study, it will be the responsibility of the anaesthesiology registrars and consultants providing the anaesthetic, to ensure patient safety and well-being, at all times. This is routine, good practise and the study will not influence or detract from these patient specific clinical decisions or patient management in any way.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving general, neuraxial, regional or local/topical anaesthesia for elective surgical intervention
* >18 years of age

Exclusion Criteria:

* Obstetric patients
* Cardiac patients

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Study Population & Sample Size:
  The study population will involve patients presenting for elective surgery, who fulfil inclusion criteria, in all surgical disciplines with elective surgical slates in the main theatre complex, during the period of the study.
  Inclusion Criteria:
  Patients included in the study will be:
  * > 18 years of age
  * Non-cardiac patients
  * Non-obstetric patients
  * Patients receiving general, neuraxial, regional or local/topical anaesthesia for elective surgical intervention
Sampling Method: Non-Probability Sample
Enrollment: 382 (Actual)
Dates: Start 2016-10-24 (Actual); Primary Completion 2016-10-31 (Actual); Study Completion 2016-10-31 (Actual)

PRIMARY OUTCOMES:
Identification and categorisation of the prevalance of hypertensive disease in adult patients presenting for non-cardiac surgery, non-obstetric elective surgery at seven hospitals in the Western Cape, South Africa. | 1 Week
  Prevalence and degree of hypertensive disease will be determined in adult patients presenting for non-cardiac, non-obstetric, elective surgery in all surgical disciplines with elective theatre lists over the period of the study at seven hospital in the Western Cape, South Africa. Serial preoperative blood pressure measurements will be performed in the pre-assessment anaesthetic consultation and in the immediate preoperative period, using an automated oscillometric blood pressure measurement technique.

CONTACTS AND LOCATIONS:
Overall Officials: Marcin Netjhardt, MMed, Principal Investigator — University of Cape Town; Francois Roodt, MMed, Study Chair — University of Cape Town; Karen van der Spuy, MBChB, Study Chair — University of Cape Town; Bruce Biccard, PhD, Study Chair — University of Cape Town; Marcelle Crowther, MBChB, Study Chair — University of Cape Town
Locations (7):
- South Africa (7):
  - Groote Schuur Hospital, Cape Town, Western Cape
  - Mitchells Plain Hospital, Cape Town, Western Cape
  - Somerset Hospital, Cape Town, Western Cape
  - Victoria Hospital, Cape Town, Western Cape
  - George Hospital, George, Western Cape
  - Paarl Hospital, Paarl, Western Cape
  - Worcester Hospital, Worcester, Western Cape

IPD SHARING:
Plan to Share IPD: Yes
Individual anonymous participant data will be collected and stored on REDCap which is a mature, secure web application for building and managing online surveys and databases. Access to individual patient information will be possible by contacting Dr MB Nejthardt at mb.nejthardt@uct.ac.za. A review of the enquiry will be undertaken by the HASS research team and the requesting person notified my email.